CLINICAL TRIAL: NCT06514365
Title: Comparison of the Analgesic Effect of Subsartorial Saphenous Block and Popliteal Sciatic vs Subsartorial Saphenous Block and IPACK in Total Knee Replacement Surgery. A Double Blind Randomized Clinical Trial.
Brief Title: Comparison of the Analgesic Effect of Subsartorial Saphenous Block and Popliteal Sciatic vs Subsartorial Saphenous Block and IPACK in Total Knee Replacement Surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Dinu, Principal Investigator, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IPACK-20
Record Dates: First submitted 2020-07-22; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Pain, Acute; Knee Osteoarthritis; Anesthesia
Keywords: Ipack; Block; Total knee replacement
MeSH Terms: conditions — Acute Pain; Osteoarthritis, Knee; Bites and Stings | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Echo-guided IPACK block (Experimental): IPACK block using 0.25% bupivacaine 15mL with adrenaline once.
  Interventions: Drug: IPACK block with Bupivacaine 0.25% with adrenaline
- Echo-guided sciatic block (Active Comparator): Sciatic nerve block using 0.25% bupivacaine 15mL with adrenaline once.
  Interventions: Drug: IPACK block with Bupivacaine 0.25% with adrenaline

INTERVENTIONS:
Drug: IPACK block with Bupivacaine 0.25% with adrenaline — The iPACK in performed in the popliteal fossa about 1 finger breath above the patella, ecoguided. That aims to anesthetize the articular branches to the posterior aspect of the knee in the popliteal region.
  Other Names: Interspace between the Popliteal Artery and the Capsule of the posterior Knee

SUMMARY:
Total knee replacement surgery is associated with significant pain in the immediate postoperative period, especially in movement. In turn, this is associated with more subsequent chronic pain.

There are multiple options and the tendency is to perform increasingly distal nerve blocks to minimize limb weakness and thus allow early rehabilitation. In 2012, in an oral communication, Sanjay Sinha described a new nerve block called iPACK ("Interspace between the Popliteal Artery and the Capsule of the posterior Knee"). There are few studies on the efficacy of such a blockade so far, but none comparing the groups saphene + sciatic blocks vs. saphene + iPACK blocks.

Therefore, this study aims to provide more information on the effectiveness this nerve blocks, in total knee replacement, in terms of analgesia and motor function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis scheduled for total primary knee arthroplasty with same surgeons
* Locoregional anesthesia
* Age equal to or greater than 18 years
* Consent to participate in the study

Exclusion Criteria:

* Age under 18 years old
* General anesthesia
* Allergy to local anesthetics
* Severe kidney failure (Cr ≥ 2mg / dL)
* Chronic opioid use (over 3 months)
* Chronic pregabalin / gabapentin use (more than 3 months)
* Psychiatric illness that may interfere with the evaluation or follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Pain at rest | 6 hours after surgery
  Measured by the numerical visual scale at 6 hours after intradural anesthesia, minimum of 0 and maximum of 10, where means no pain and 10 means the worst pain in the life of the patient.
Pain at rest | 24 hours after surgery
  Measured by the numerical visual scale at 24 hours after intradural anesthesia, minimum of 0 and maximum of 10, where means no pain and 10 means the worst pain in the life of the patient.
Pain at rest | 48 hours after surgery
  Measured by the numerical visual scale at 48 hours after intradural anesthesia, minimum of 0 and maximum of 10, where means no pain and 10 means the worst pain in the life of the patient.
Pain at movement | 6 hours after surgery
  Measured by the numerical visual scale at 48 hours after intradural anesthesia, minimum of 0 and maximum of 10, where means no pain and 10 means the worst pain in the life of the patient.
Pain with movement | 24 hours after surgery
  Measured by the numerical visual scale at 48 hours after intradural anesthesia, minimum of 0 and maximum of 10, where means no pain and 10 means the worst pain in the life of the patient.
Pain with movement | 48 hours after surgery
  Measured by the numerical visual scale at 48 hours after intradural anesthesia, minimum of 0 and maximum of 10, where means no pain and 10 means the worst pain in the life of the patient.
Motor block | 6 hours after surgery
  Measured on a scale of 3, where 0 = no motor block, 1 = partial motor block and 2 = complete motor block. It will be performed on plantar flexion (distribution of the tibial nerve) and dorsiflexion (peroneal distribution)).
Motor block | 24 hours after surgery
  Measured on a scale of 3, where 0 = no motor block, 1 = partial motor block and 2 = complete motor block. It will be performed on plantar flexion (distribution of the tibial nerve) and dorsiflexion (peroneal distribution)).
Motor block | 48 hours after surgery
  Measured on a scale of 3, where 0 = no motor block, 1 = partial motor block and 2 = complete motor block. It will be performed on plantar flexion (distribution of the tibial nerve) and dorsiflexion (peroneal distribution)).

SECONDARY OUTCOMES:
Opioids dose | 6 hours after surgery
  Measured in milligrams of intravenous morphine hydrochloride daily.
Opioids dose | 24 hours after surgery
  Measured in milligrams of intravenous morphine hydrochloride daily.
Opioids dose | 48 hours after surgery
  Measured in milligrams of intravenous morphine hydrochloride daily.
Discharge days | Days
  Time to discharge measured in days
Patient satisfaction | 24 hours after surgery
  Patient satisfaction on a scale of 0 to 10, where 0 is minimum satisfaction and 10 is maximum satisfaction.
Ambulation time | Up to 24 hours
  Time to ambulation (measured in hours) from discharge from URPA

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No